CLINICAL TRIAL: NCT01925534
Title: Pilot Study of Optiflow as a NIV Rest Therapy
Brief Title: Pilot Study of High-flow Humidified Nasal Oxygen During Breaks From Noninvasive Ventilation
Acronym: OPTINIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FPH-OF13-01; IRB-10967 (Other: IRB Tufts Medical Center)
Record Dates: First submitted 2013-07-31; First posted 2013-08-19 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Acute Respiratory Failure; Treatment With Noninvasive Positive Pressure Ventilation
Keywords: Optiflow; Humidified high-flow oxygen therapy; Noninvasive ventilation; Acute respiratory failure; Standard oxygen therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optiflow (Experimental): High-flow humidified nasal oxygen delivery system
  Interventions: Device: High-flow humidified nasal oxygen delivery system
- Oxygen therapy (Active Comparator): Standard oxygen therapy
  Interventions: Device: Standard oxygen therapy

INTERVENTIONS:
Device: High-flow humidified nasal oxygen delivery system — During breaks from NIV oxygen will be provided through the Optiflow with FiO2 and flow-rate titrated to maintain the oxygen saturation (SpO2) above 90%.
  Other Names: Optiflow
  Arms: Optiflow
Device: Standard oxygen therapy — During breaks from NIV oxygen will be provided by standard nasal cannula or mask to maintain the SpO2 above 90%.
  Arms: Oxygen therapy

SUMMARY:
The purpose of this study is to assess whether Optiflow, a high-flow humidified oxygen delivery system, is superior to standard oxygen therapy during breaks off noninvasive ventilation in patients affected by acute respiratory failure and in respiratory distress. The investigators anticipate that the Optiflow will provide oxygen more effectively, be more comfortable and permit longer breaks off NIV, shortening the total duration of NIV.

DETAILED DESCRIPTION:
Background: Noninvasive ventilation (NIV) provides respiratory support to many patients affected by acute respiratory failure. This treatment, compared to invasive mechanical ventilation, allows patients to take intermittent breaks during which oxygen therapy is provided through a nasal cannula or mask. During these breaks, the lack of ventilator support may predispose to respiratory distress, retention of CO2 and oxygen desaturation. Optiflow is a nasal humidified (37◦C, 44mg/L H2O) high-flow (up to 60 L/min) therapy which can provide greater support than standard oxygen therapy during the breaks from NIV.

Aim of the study is to evaluate Optiflow as an alternative to standard oxygen therapy during breaks from NIV in patients with acute respiratory failure. The investigators hypothesize tha Optiflow will reduce the total length of stay on NIV, and increase the comfort and length of the breaks. Also, the investigators anticipate that it will reduce respiratory rate, accessory muscle use and dyspnea score compared to standard oxygen therapy.

Experimental design Prospective open-label, parallel, randomized (1:1) controlled study, with a target enrollment of 70.

Study procedures Enrolled patients receiving NIV will be randomized into two arms; a treatment group which will receive Optiflow during breaks and a control arm which will receive standard oxygen therapy during breaks. In both cases, FiO2 will be titrated to maintain oxygen saturation above 90%. The necessity of breaks will be determined together with the patients (talk, eat, medication, communicate with family, inability to tolerate the interface), and the need to resume NIV will be based on clinical data, such as dyspnea, respiratory rate, heart rate, blood pressure, oxygen saturation, transcutaneous carbon dioxide (CO2) and patients' desire.

Recorded data: The investigators will record demographic baseline data; Glasgow Coma Scale, respiratory and heart rate, blood pressure, dyspnea score, accessory muscle use, and comfort score at randomization, at the end of each NIV session and NIV break; the length of each NIV session and break; the medications administered and all the arterial blood gases (ABG) on a daily basis. Moreover the investigators will record the NIV parameters and inspired oxygen fraction (FiO2) at each session and break.

Risks: The investigators don't anticipate any significant risks related to the study procedures and equipment. Some patients may not tolerate the Optiflow and some patients may fail NIV and require intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 or more years of age treated with Bipap or CPAP as per hospital protocol, with an underlying clinical diagnosis of acute respiratory failure.
* Patients that, prior to administration of NIV, had persistent respiratory acidosis with a pH <7.35 and arterial CO2 > 45 mmHg despite controlled oxygen therapy and standard medical management i.e. bronchodilators, corticosteroids and antibiotics, or
* Patients with hypoxemic respiratory failure with a PaO2/FiO2 ratio < 300 and respiratory rate ≥ 24.
* Anticipated duration on NIV of at least 24 hrs

Exclusion criteria:

* Usual contraindications to NIV
* Respiratory arrest
* Unable to fit mask
* Medically unstable or multiple organ failure or unstable coronary disease
* Agitated or uncooperative
* Unable to protect airways
* Swallowing difficulties
* Excessive secretions not managed by clearance techniques
* Recent upper airway or gastro-intestinal surgery
* Facial deformity or previous head and neck surgery
* Undrained pneumothorax
* NIV failure within first 2 hours (either intolerance or requirement for intubation)
* Managed for greater than 48 hours on NIV prior to randomization
* Disorientation, confusion, unable to rate comfort or dyspnea
* Expected to require NIV for fewer than 24 hrs from the time of enrollment
* Patient previously in study
* Patients on CPAP nighttime only due to OSA

Withdrawal/Termination criteria:

* Patients will be withdrawn from the study when NIV fails and/or the patient is intubated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Hill, MD, Principal Investigator — Tufts Medical Center
Locations (2):
- United States (2):
  - Intensive Care Unit and Intermediate Care Unit, Tufts Medical Center, Boston, Massachusetts
  - Intensive Care Unit, Winchester Hospital, Winchester, Massachusetts

REFERENCES:
- [Background] Ricard JD, Boyer A. Humidification during oxygen therapy and non-invasive ventilation: do we need some and how much? Intensive Care Med. 2009 Jun;35(6):963-5. doi: 10.1007/s00134-009-1457-9. Epub 2009 Mar 18. No abstract available. PMID 19294364
- [Background] El-Khatib MF. High-flow nasal cannula oxygen therapy during hypoxemic respiratory failure. Respir Care. 2012 Oct;57(10):1696-8. doi: 10.4187/respcare.02072. No abstract available. PMID 23013907
- [Background] Sztrymf B, Messika J, Bertrand F, Hurel D, Leon R, Dreyfuss D, Ricard JD. Beneficial effects of humidified high flow nasal oxygen in critical care patients: a prospective pilot study. Intensive Care Med. 2011 Nov;37(11):1780-6. doi: 10.1007/s00134-011-2354-6. Epub 2011 Sep 27. PMID 21946925
- [Background] Roca O, Riera J, Torres F, Masclans JR. High-flow oxygen therapy in acute respiratory failure. Respir Care. 2010 Apr;55(4):408-13. PMID 20406507
- [Background] Parke RL, Eccleston ML, McGuinness SP. The effects of flow on airway pressure during nasal high-flow oxygen therapy. Respir Care. 2011 Aug;56(8):1151-5. doi: 10.4187/respcare.01106. Epub 2011 Apr 15. PMID 21496369
- [Background] Corley A, Caruana LR, Barnett AG, Tronstad O, Fraser JF. Oxygen delivery through high-flow nasal cannulae increase end-expiratory lung volume and reduce respiratory rate in post-cardiac surgical patients. Br J Anaesth. 2011 Dec;107(6):998-1004. doi: 10.1093/bja/aer265. Epub 2011 Sep 9. PMID 21908497
- [Background] Parke RL, McGuinness SP, Eccleston ML. A preliminary randomized controlled trial to assess effectiveness of nasal high-flow oxygen in intensive care patients. Respir Care. 2011 Mar;56(3):265-70. doi: 10.4187/respcare.00801. Epub 2011 Jan 21. PMID 21255498
- [Background] Braunlich J, Beyer D, Mai D, Hammerschmidt S, Seyfarth HJ, Wirtz H. Effects of nasal high flow on ventilation in volunteers, COPD and idiopathic pulmonary fibrosis patients. Respiration. 2013;85(4):319-25. doi: 10.1159/000342027. Epub 2012 Nov 1. PMID 23128844

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Optiflow | Oxygen Therapy
Started | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Optiflow | Oxygen Therapy | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (13.8) | 63.4 (14.0) | 66.17 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay on Noninvasive Ventilation (NIV)
Description: The investigator will measure the total time on NIV in day(s), hours and minutes. This is done by having nursing staff note times of NIV start to finish of each session of NIV. They were added to get cumulative time.
Time Frame: Day 1-7
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Optiflow | Oxygen Therapy
Number analyzed (Participants) | 23 | 24
Minutes | 1404 (1386) | 1386 (951)

2. Secondary Outcome: Length of Breaks From NIV
Description: This is done by having nursing staff note times of break start (off NIV) to start of next session of NIV in minutes. Subgroup analysis was performed to assess differences between hypercapnic and hypoxemic patients, not observed in terms of time spent on or off NIV.
Time Frame: Day 4-10
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Optiflow | Oxygen Therapy
Number analyzed (Participants) | 23 | 24
minutes | 1345 (902) | 1221 (770)

3. Secondary Outcome: Assessment of Respiratory Rate During Break
Description: Evaluation of respiratory rate. This was counted for a minute at bedside at start and finish of break.
Time Frame: day 1-4
Population: Two groups randomly allocated to High Flow or Standard oxygen therapy
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Optiflow | Oxygen Therapy
Number analyzed (Participants) | 23 | 24
breaths/min
  Respiratory Rate: Break | 23.8 (6.8) | 21.8 (5.2)
  Respiratory Rate: NIV | 23.3 (5.3) | 20.1 (4.1)

4. Secondary Outcome: Patients' Comfort
Description: Using a visual analogue scale (VAS). Patients rate how comfortable they felt on a 1 to 10 scale with 10 being most comfortable and 1 being the least comfortable.
Time Frame: Day 2-4
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Oxygen: Standard oxygen therapy
  Standard oxygen therapy: During breaks from NIV oxygen will be provided by standard nasal cannula or mask to maintain the SpO2 above 90%.
Arm/Group | Optiflow | Oxygen
Number analyzed (Participants) | 23 | 24
score on a scale
  VAS Comfort Score Break | 8.3 (2.7) | 6.9 (2.3)
  VAS Comfort Score NIV | 5.9 (3.9) | 6.2 (2.9)

5. Secondary Outcome: Oxygen Saturation During Breaks
Description: Using pulse oximetry (SpO2) at beginning and end of breaks
Time Frame: day 1-4
Measure: Mean (Standard Deviation); unit: arterial oxygen saturation (%)
Arm/Group | Optiflow | Oxygen Therapy
Number analyzed (Participants) | 23 | 24
arterial oxygen saturation (%)
  SpO2, % mean: Break | 94.1 (3.2) | 94.7 (2.1)
  SpO2, % final: Break | 93.7 (5.0) | 95.4 (2.7)
  SpO2, % final: NIV | 95.9 (2.9) | 96.4 (2.0)

6. Secondary Outcome: Need for Intubation
Description: Count of participants who underwent endotracheal intubation
Time Frame: Days 2-10
Measure: Count of Participants; unit: Participants
Arm/Group | Optiflow | Oxygen Therapy
Number analyzed (Participants) | 23 | 24
Participants | 2 | 0

7. Secondary Outcome: Ease of Eating
Description: difficulty eating using patient rating on a visual analog scale of 0 for easy eating and 4 for difficult eating. Results tabulated as number of patients finding it easy to eat (Score of 0-1)
Time Frame: Day 1-4
Measure: Count of Participants; unit: Participants
Arm/Group | Optiflow | Oxygen Therapy
Number analyzed (Participants) | 23 | 24
Participants | 20 | 15

ADVERSE EVENTS:
Arm/Group | Optiflow | Oxygen Therapy
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/23 | 0/24
Other Adverse Events (participants affected / at risk) | 11/23 | 15/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optiflow (N=23) | Oxygen Therapy (N=24)
endotracheal intubation (ETI) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optiflow (N=23) | Oxygen Therapy (N=24)
Nasal Dryness (Ear and labyrinth disorders) | 11 (11) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No